CLINICAL TRIAL: NCT06093074
Title: Self-management Program for Patients in the Sub-acute Phase After Moderate to Severe Traumatic Injury -a Feasibility Study
Brief Title: Self-management Program for Patients in the Sub-acute Phase After Traumatic Injury - a Feasibility Study
Acronym: SMS_trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sunnaas Rehabilitation Hospital (Other); South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Nada Andelic, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: msrasmussen
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Self-management; Feasibility Studies; Spinal Cord Injuries; Brain Injuries
Keywords: traumatic injuries; multi trauma; interventions
MeSH Terms: conditions — Spinal Cord Injuries; Brain Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a feasibility trial evaluating the feasibility and acceptability of a planned randomized controlled trial. Therefore, no control group will be included in this feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): Feasibility trial study group.
  Interventions: Behavioral: self-management program after traumatic injuries

INTERVENTIONS:
Behavioral: self-management program after traumatic injuries — The self-management support (SMS) program is manualized and will include eight weekly 2.5-hour sessions in groups of 5-7 participants. This feasibility trial will assess both face-to-face delivered program and a tele-health program via electronic devices. The tele-health intervention will be delivered with the same SMS content, frequency, and in-group mode.

SUMMARY:
The goal of this descriptive non-randomized feasibility study is to assess aspects of feasibility of the intervention arm in a planned full-scale randomized controlled trial testing the effectiveness of a self-management program for persons who have sustained a moderate to severe traumatic injury. All outcomes will be evaluated based on pre-defined success criteria. The main outcomes in the feasibility study are:

* Consent rate of eligible patients
* Drop-out rate
* Attendance rate in the program sessions

Secondary outcomes are the participants' acceptance, reception, and perceived usefulness. Other outcomes are fidelity and protocol adherence, as well as the feasibility of a telehealth version of the program and the data collection methods.

The participants will receive a group-based self-management program consisting of eight weekly 2.5-hour sessions delivered by a multidisciplinary team. The self-management program is manualized and includes psychoeducation, training in self-management skills and strategies, setting goals, action planning, and sharing of experiences. The participants will also complete the pre- and post-intervention assessments.

DETAILED DESCRIPTION:
Background: Traumatic injuries, defined as physical injuries with sudden onset, are a major cause of distress and disability, with far-reaching societal consequences. A significant proportion of trauma survivors report problems and impaired health years after the injury. This includes impaired physical and mental health, difficulties in daily activities, and reduced health-related quality of life, which may subsequently limit participation in work/study, leisure activities, and family life. Consequently, these patients are often in need of complex rehabilitation and long-term follow-ups. The need to improve rehabilitation services and provision, including shared decision-making and self-management approaches, has been acknowledged. The World Health Organisation's (WHO) Rehabilitation 2030 initiative calls for strengthening and developing multidisciplinary rehabilitation. In line with the principles of user-involvement and patient-centred rehabilitation, strategies aiming to support self-management have received increased attention. Self-management refers to the systematic provision of education and supportive interventions by health care staff to increase patients' skills and confidence in managing their health problems. As recommended by the complex intervention framework presented by the Medical Research Council (MRC), a feasibility study will be performed as a preparation of a randomized controlled trial (RCT) on the effectiveness of a self-management support program.

Design and study settings: a non-randomized feasibility study of the intervention arm performed as a preparation for a pragmatic RCT testing the effectiveness of a self-management program using a mixed-methods design with 6-months follow-up. The feasibility study will be conducted at Oslo University Hospital and eligible patients who have sustained a moderate to severe traumatic injury will be included 3-4 months post-injury. Informed consent will be collected.

Intervention: The self-management program is manualized and integrates components from evidence-based rehabilitation strategies within relevant functional domains, to fit the symptom burden of the trauma population. It consists of eight 2-5-hour sessions delivered by a multidisciplinary team. The program will be delivered both face-to-face and in a telehealth version and patients will choose the delivery format based on their own preferences.

Aim: The overall aim is to set up the program, make necessary adjustment of the program, and study procedures in advance of the full-scale RCT. More specifically, feasibility of the intervention program and study procedures (including acceptability, protocol adherence, consent rates, dropout, attendance rate, participants' satisfaction with the program, and data collection methods) will be assessed.

Sample size and analyses: In the feasibility study, 10% of the estimated sample size in the intervention arm of the full-scale RCT will be included, which equals to 12 participants. The results will be evaluated according to pre-defined success criteria to determine feasibility and make necessary adjustments to the SMS program and study procedures in advance of the full-scale RCT.

To describe the study population, the following sociodemographic and injury-related variables will be recorded at baseline: age, gender, marital status, living conditions, educational level, description of pre-injury functioning and employment. Medical variables include comorbidities, diverse injury characteristics and trauma severity scores, length of hospitalisation and medical treatment modalities, and symptom burden along with screening of cognitive function.

Data collection methods and completion of the selected outcome measures will be assessed in the feasibility study. The following outcome measures are planned for the full-scale RCT, and will also be included in the feasibility study:

* Self-efficacy assessed using the Trauma Coping Self-Efficacy questionnaire
* Symptom burden assessed by the Rivermead Post-Concussion Symptom Questionnaire, Fatigue Severity Scale, Insomnia Severity Index, and Brief Pain Inventory Short Form
* Physical function assessed by the Short Physical Performance Battery and the International Physical Activity Questionnaire Short Form
* Cognitive function assessed by the Cognitive Failures Questionnaire and Cognitive items Rivermead.
* Emotional distress assessed by the Patient Health Questionnaire-9 & Generalized Anxiety Disorder-7 and Impact of Event Scale- Revised
* Return to work assessed by the full-time/part-time (percentage) or hours per week working
* Resilience assessed by the Resilience Scale for Adults
* Health status assessed by EuroQol five-dimensional questionnaire
* Individual injury related self-reported problem areas assessed by the target outcomes
* Evaluation of changes and intervention satisfaction assessed by the Patient Global Impression of Change and Visual Analogue Scales
* Disability assessed by the WHO Disability Assessment Scale
* General functioning assessed by the Glasgow Outcome Scale - Extended.
* Communication assessed by Communication with physicians and Health Literacy Questionnaire
* Health care utilization assessed by the type and frequency of health care services received

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18-72 years residing in the southeast region of Norway
2. Admitted to OUH directly or after transfer from local hospitals within 72 hours of injury
3. At least a two-day hospital stay
4. Traumatic injury corresponding to a New Injury Severity Scale score (NISS) >9
5. Patients reporting injury-related symptoms, functional impairments, and/or difficulties with daily activities at discharge from Oslo University Hospital
6. Time since injury 3-4 months post-injury at inclusion.

Exclusion Criteria:

1. Cognitive function corresponding to a Mini Mental Status score <20 points
2. Severe psychiatric diseases or drug/alcohol dependence that require treatment
3. Complete spinal cord injury or isolated abdominal/thoracic injuries
4. Insufficient command of Norwegian.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Consent rate of eligible | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Recruitment procedures will be assessed by consent rate.
  Highly feasible: More than 75-100 % consent rate Moderately feasible: 50-74% consent rate Not feasible: Less than 50% consent rate
Drop-out rate | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Recruitment procedures will be assessed by drop-out rate.
  Highly feasible: Less than 25% drop-outs Moderately feasible: 35-26% drop-outs Not feasible: More than 35% drop-outs
Attendance rate | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Acceptability for participants will be assessed by percentage of sessions attended.
  Highly feasible: 90% or more attendance Moderately feasible: 75%-89% attendance Not feasible: Less than 75% attendance

SECONDARY OUTCOMES:
Patient acceptability and receipt | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Acceptability for participants and therapist will be assessed by patient acceptability and receipt rated by therapist checklist. This scale is rated on a Likert scale from 0 to 3.
  Highly feasible: Mean score 2 or above Moderately feasible: Mean score between 1 and 2 Not feasible: Mean score lower than 1
Usefulness of intervention rated by participants | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Usefulness of intervention rated by participants will be assessed by rating of each session on a Likert scale from 1 (not useful) to 5 (extremely useful). The total mean score of the scale will determine the perceived usefulness of each session (from session 1 to session 8).
  Highly feasible: Mean score of 4 or above ("very useful" to "extremely useful) Moderately feasible: Mean score between 2 ("somewhat useful") and 3 ("moderately useful") Not feasible: Mean score lower than 2 ("not useful")
Recommendation to others | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Usefulness of intervention rated by participants by answering question wether or not they would recommend program to others (yes or no).
  Highly feasible: 80% or more positive to recommend program to others. Moderately feasible: 65-79% positive to recommend program. Not feasible: Less than 65% positive to recommend program.

OTHER OUTCOMES:
Fidelity of therapists' adherence | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Quality of the treatment delivery will be assessed by fidelity monitoring of therapists' adherence and competency in delivering program content will be assessed by senior investigators rating of fidelity checklist, rated on a Likert scale from 0 (poor) to 2 (excellent).The fidelity checklist total mean score will determine the fidelity.
  Highly feasible: Mean score 2 ("excellent") Moderately feasible: Mean score 1 ("good") Not feasible: Mean score 0 ("poor")
Protocol adherence by study-specific checklists. | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Quality of the treatment delivery will be assess by therapists monitoring the discrepancies between intervention delivery and the intervention manual by using extensive checklists relating to each of the intervention sessions. The number of non-delivered treatment components will be counted, and the percentage of deviation will be calculated compared to the total number of intervention components per session.
  Highly feasible: Less than 15% deviation Moderately feasible: 16-25% deviation Not feasible: More than 25% deviation
Feasibility of telehealth intervention by technical log over reported technical failures (by therapist). | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Quality of the treatment delivery will be assessed by the feasibility of telehealth intervention. Therapist-recorded technical failures in using telehealth platform for intervention delivery will be used, where therapists record in a technical log the number of sessions interrupted due to technical failures per session.
  Highly feasible: Restart of equipment in 0-1 session per group Moderately feasible: Restart in 2-3 sessions per group Not feasible: Restart in more than 4 sessions per group
Duration of baseline assessment | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Evaluation of methods and assessment at baseline will be assessed by duration of the baseline assessment.
  Highly feasible: Less than 2 h. Moderately feasible: 2-3 h. Not feasible: More than 3 h.
Duration of T2 (follow-up at end of intervention) | Will be evaluated after the intervention period, i.e. 2-3 months after inclusion
  Evaluation of methods and assessment at the follow-up will be assessed by duration of the follow-up at the end of intervention.
  Highly feasible: Less than 2 h. Moderately feasible: 2-3 h. Not feasible: More than 3 h.

CONTACTS AND LOCATIONS:
Overall Officials: Nada Andelic, Phd, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data are sensitive and will not be openly shared.

REFERENCES:
- [Background] Bonatti H, Calland JF. Trauma. Emerg Med Clin North Am. 2008 Aug;26(3):625-48, vii. doi: 10.1016/j.emc.2008.05.001. PMID 18655938
- [Background] Gabbe BJ, Simpson PM, Cameron PA, Ponsford J, Lyons RA, Collie A, Fitzgerald M, Judson R, Teague WJ, Braaf S, Nunn A, Ameratunga S, Harrison JE. Long-term health status and trajectories of seriously injured patients: A population-based longitudinal study. PLoS Med. 2017 Jul 5;14(7):e1002322. doi: 10.1371/journal.pmed.1002322. eCollection 2017 Jul. PMID 28678814
- [Background] Geraerds AJLM, Richardson A, Haagsma J, Derrett S, Polinder S. A systematic review of studies measuring health-related quality of life of general injury populations: update 2010-2018. Health Qual Life Outcomes. 2020 May 29;18(1):160. doi: 10.1186/s12955-020-01412-1. PMID 32471430
- [Background] Huang S, Dipnall JF, Gabbe BJ, Giummarra MJ. Pain and mental health symptom patterns and treatment trajectories following road trauma: a registry-based cohort study. Disabil Rehabil. 2022 Dec;44(25):8029-8041. doi: 10.1080/09638288.2021.2008526. Epub 2021 Dec 6. PMID 34871122
- [Background] World Health Organization. Rehabilitation 2030 Initiative. 2017 [cited 2022 29.07.22]; Available from: https://www.who.int/initiatives/rehabilitation-2030.
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Sohlberg, M.M., Cognitive Rehabilitation Manual: Translating Evidence-Based Recommendations into Practice. Archives of clinical neuropsychology, 2012. 27(8): p. 931-932.
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Benight CC, Shoji K, James LE, Waldrep EE, Delahanty DL, Cieslak R. Trauma Coping Self-Efficacy: A Context-Specific Self-Efficacy Measure for Traumatic Stress. Psychol Trauma. 2015 Nov;7(6):591-599. doi: 10.1037/tra0000045. PMID 26524542